CLINICAL TRIAL: NCT04792281
Title: Impact of FDG-PET/CT on Management of Patients with Native Valve Infective Endocarditis
Acronym: PET-NAVIE
Status: Recruiting | Type: Observational
Sponsor: Montreal Heart Institute (Other)
Responsible Party: Principal Investigator, Matthieu Pelletier-Galarneau, MD MSc, Assistant Professor, Montreal Heart Institute
Other Study IDs: MP-33-2020-2674
Record Dates: First submitted 2021-03-05; First posted 2021-03-10 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Infective Endocarditis; Native Valve Endocarditis
Keywords: PET/CT; FDG; Duke Criteria
MeSH Terms: conditions — Endocarditis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with suspected native valve endocarditis

SUMMARY:
The proposed study is a multicentric prospective observational cohort study of patients with suspected NVE. The study population includes those with Possible IE according to the modified Duke criteria and investigated at one of the 6 participating sites which include 2 cardiac centers, the MHI and the IUCPQ, as well as 4 tertiary care centers, the Jewish General Hospital , the McGill University Health Centre and the CHUS.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older, capable to provide informed consent;
* Referred for a FDG-PET/CT study
* Classified as having Possible IE prior to FDG-PET/CT imaging;
* Patients must be able to tolerate the physical/logistical requirements of a PET/CT scan.

Exclusion Criteria:

* Subjects with prosthetic cardiac valve and/or CIED;
* Pregnant or breastfeeding female;
* Body mass index > 45 kg/m2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes those with Possible IE according to the modified Duke criteria and investigated at one of the 5 participating sites
Sampling Method: Non-Probability Sample
Enrollment: 97 (Estimated)
Dates: Start 2021-08-31 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with Possible IE that will be appropriately reclassified | 3 months
  Proportion of patients with Possible IE that will be appropriately reclassified as Definite IE by the addition of FDG-PET to the Duke criteria.

SECONDARY OUTCOMES:
Sensitivity, specificity, and accuracy of FDG-PET for the detection of NVE | 3 months
Sensitivity, specificity, and accuracy of the Duke criteria with FDG-PET for detection of NVESensitivity, specificity, and accuracy of the Duke criteria with FDG-PET for detection of NVE | 3 months
Sensitivity, specificity, and accuracy of the Duke criteria with FDG-PET but excluding TEE for the detection of NVE | 3 months
Differences in maximal standardized uptake value (SUVmax) between infected and non-infected valves | 3 months
Differences target-to-background ratio (TBR) between infected and non-infected valves | 3 months
Proportion of patients in whom a TEE was not necessary to diagnose NVE through the addition of FDG-PET | 3 months
Proportion of patients with final diagnosis of IE with septic emboli detected on whole body FDGPET | 3 months
Differences in the rate of sub-optimal suppression protocol between males and females | 3 months
Proportion of patients with incidental cancer identified on FDG-PET | 3 months

OTHER OUTCOMES:
Correlation between the diagnostic accuracy and available demographic, technical, and clinical factors | 3 months
  Correlation between the diagnostic accuracy (false-negative/false-positive studies versus truenegative/true-positive) and the available demographic and clinical factors (age, sex, duration of antibiotherapy, blood glucose, CRP, history of renal failure, history of malignancy, history of diabetes, chronic liver disease, time since onset of symptoms, and quality of myocardial suppression) as well as camera system (analog vs digital)
Difference in the area under the curve (c-statistic) of the Duke criteria with TEE but excluding FDG-PET, with TEE and FDG-PET, and with FDG-PET but excluding TEE | 3 months
Differences in sensitivity, specificity, and accuracy of FDG-PET with and without respiratory and ECG-gated acquisitions | 3 months

CONTACTS AND LOCATIONS:
Locations (6):
- Canada (6):
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - Montreal Heart Institute, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - McGill University Health Center, Montreal, Quebec
  - University Institute of Cardiology and Respirology of Quebec, Québec, Quebec
  - Centre Hospitalier de l'Universite de Sherbrooke, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: Undecided